CLINICAL TRIAL: NCT03582150
Title: Ambulatory Alcohol Detoxification With Remote Monitoring
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding lost during COVID
Sponsor: Stanford University (Other)
Collaborators: SoberLink, LLC (Industry)
Responsible Party: Principal Investigator, Anna Lembke, Clinical Associate Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-44681
Record Dates: First submitted 2018-06-27; First posted 2018-07-10 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Alcohol Use Disorder
Keywords: Ambulatory alcohol detoxification; alcohol withdrawal; remote monitoring with breathalyzer
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Receiving Soberlink Device (Experimental)
  Interventions: Device: Remote Monitoring with Ambulatory Detox

INTERVENTIONS:
Device: Remote Monitoring with Ambulatory Detox — * Each Subject willing to participate will sign an Informed Consent and will receive a Subject Number.
  * Study staff will assist Subject in setting up the Soberlink Device as well as the Bluetooth enabled blood pressure cuff and Smartphone APP.
  * Study staff documents Subject's resting and standing blood pressure and pulse to establish a safety range for the study.
  * Subjects will use the blood pressure cuff and the Soberlink Device four times a day per a set schedule to determine blood pressure and pulse and blood alcohol concentration (BAC). Results will be sent to the Soberlink System for study staff to review.
  * If the Subject misses a Soberlink test, tests positive for alcohol, or the identity cannot be approved, the staff will be immediately notified by the Soberlink System.
  * The Subject will be enrolled on a Monday and evaluated by the study physician and return to the site for an evaluation by the study physician and staff on Tuesday, and a final assessment on Thursday.

SUMMARY:
This study is designed to examine the feasibility and impact of the use of remote monitoring devices during an outpatient ambulatory alcohol detoxification treatment for patients with alcohol use disorders.

DETAILED DESCRIPTION:
The study will include 30 subjects with a diagnosis of alcohol use disorder. The study uses a breathalyzer device with facial recognition to confirm the patient's identity and sends the information to the study staff using cellular technology. A second device is used which is a wireless blood pressure cuff that connects to the patient's smartphone and sends blood pressure and heart rate measurements directly to the study physician for enhanced monitoring during alcohol withdrawal management. The duration of the study is 8 days, starting with an initial appointment to set up the equipment. Throughout the study, surveys are completed by subjects in regards to their experience with the device. Subjects undergo a brief 30-60 minute appointment on the first day of the study, appointments as needed throughout the study, and an appointment on the last day of the study to check in with the physician for ongoing ambulatory management of alcohol withdrawal, including medication adjustments if indicated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Subject between the ages of 21-75 years old
* Meeting DSM-V criteria for alcohol use disorder and needing medically supervised detoxification based on medical history and pattern of alcohol use delineated by timeline follow back method.
* Has 24/7 easy access to a hospital. This is to ensure easy admission to a higher level of care if indicated.
* Willing to use the Soberlink Device to provide blood alcohol concentration (BAC)
* Willing to use the blood pressure cuff to provide blood pressure and pulse (BPPT) measurement
* Willing to sign an informed consent

Exclusion Criteria:

* BAC above the legal driving limit at the time of screening
* Developing symptoms or history of symptoms of severe withdrawal syndrome such as fever, disorientation, drenching sweats, severe tachycardia, or severe hypertension
* History of delirium tremens or seizures
* Co-morbid medical or psychiatric history requiring inpatient admission for careful monitoring
* Subject unwilling to respond to redirection when blood pressure and heart rate warning signs are triggered
* Does not have an iPhone, iPod, iPad, or Apple Watch with iOS 7.0 or later, or does not have an Android phone or tablet with Android 4.4 or later
* Unable or unwilling to properly use the monitoring devices, or find the monitoring devices an obstruction to comply with treatment
* Subject that is non-English speaking
* Subject that is a child, adolescent, or cognitively impaired

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants completing the eight-day protocol using Soberlink Device | Baseline to end of study (eight days).
  The Subject will be enrolled on day one and return to the site for an evaluation by the study staff on day eight. They will be seen by study staff as needed throughout the study for withdrawal management. If Subject complies with the guidelines of the study, medications will be prescribed. On or after the last day of the study, the Subject will return to the study site for a final evaluation outcomes.

SECONDARY OUTCOMES:
Missed Soberlink test | Baseline to end of study (eight days)
  If a scheduled Soberlink test is missed, Contacts will be notified. It is encouraged that the Subject submits an unscheduled test as soon as possible. If tests are repeatedly missed, the physician on duty will make a clinical determination whether to continue treatment, modify the treatment protocol, or advise transitioning to inpatient treatment immediately.
Positive BAC test received from Soberlink | Baseline to end of study (eight days)
  If a positive BAC test is received, contacts will be notified. The Soberlink System will automatically engage the Subject in a Retest cycle. The Device screen will prompt the Subject to Retest in 15 minutes, and the Subject will receive an automated text message to their mobile phone informing them that because they submitted a positive test, they are now in a Retest cycle. If the confirmation test has a positive BAC, the Subject will be asked to Retest every 15 minutes until a compliant test is submitted, or until 3 hours have elapsed. Failing to follow the on-screen instructions and text message reminders will be considered noncompliance and a violation of the protocol.
Scheduled Blood pressure and heart rate test is missed or out of range | Baseline to end of study (eight days)
  If a scheduled test is missed, it is encouraged that the Subject submits an unscheduled test as soon as possible. If tests are repeatedly missed, the physician on duty will make a clinical determination whether to continue treatment, modify the treatment protocol, or advise transitioning to inpatient treatment immediately.
Subject's self-report on effect of breathalyzer device on their behavior | Baseline to end of study (eight days)
  Subjects will fill out surveys on the effect of using the device on their cravings and relapse.
Adverse events | Baseline to end of study (eight days)
  If Subject experiences any adverse events, the Subject should contact the study staff, or call 9-1-1. The physician on duty will make a clinical determination whether to continue treatment, modify the treatment protocol, or advise transitioning to inpatient treatment immediately.
Subject not agreeable to clinical recommendations | Baseline to end of study (eight days)
  If the Subjects are not agreeable to clinical recommendations, treatment will be discontinued and considered against advice. The Subject will be removed from the study, and no further clinical action will be taken. The Subject can always reconsider and return to the hospital for review of appropriate level of care.

CONTACTS AND LOCATIONS:
Overall Officials: Amer Raheemullah, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Addiction Medicine and Dual Diagnosis Clinic, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No